CLINICAL TRIAL: NCT07011615
Title: Feasibility/Acceptability of a Brief Motivational Intervention Integrating Online Personalized Feedback & Tailored Text Messages for Frequent/High-Intensity Cannabis Use in Post-Legalization Landscape
Brief Title: Feasibility/Acceptability of a Brief Motivational Intervention for Frequent/High-Intensity Cannabis Use
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Christine Lee, Research Professor, School of Medicine: Psychiatry, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00020546; 1R34DA061049-01 (NIH)
Record Dates: First submitted 2025-06-05; First posted 2025-06-09 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Cannabis Use
MeSH Terms: interventions — Telemedicine; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Motivational Mobile Health (mHealth) Intervention (Experimental): Participants randomized to the Brief Motivational mHealth intervention will experience a five week self-directed web-based intervention with text messages.
  Interventions: Behavioral: Brief Motivational Mobile Health (mHealth) Intervention
- Psychoeducational Attention Control (Other): Participants randomized to the control group will receive a program to learn more about psychoeducational information about cannabis. They will receive psychoeducational material via text messages.
  Interventions: Other: Psychoeducational Attention Control (AC)

INTERVENTIONS:
Behavioral: Brief Motivational Mobile Health (mHealth) Intervention — Participants randomized to the mHealth intervention condition will receive a five-week online program that incorporates weekly text messages. The program will begin with prompting the young adult to reflect on their journey with cannabis and to reflect on their personal goals and how cannabis is reflected in these goals and how their social network may support their goals. Additional mini-modules are included related to topics such as motivations for use, perceived norms and tracking cannabis use. Text messages will be sent weekly to return to the program to prompt reflection and support any goals the participant indicates.
  Arms: Brief Motivational Mobile Health (mHealth) Intervention
Other: Psychoeducational Attention Control (AC) — Participants randomized to the control group will receive a program to learn more about psychoeducational information about cannabis. They also receive psychoeducational material via text messages.
  Arms: Psychoeducational Attention Control

SUMMARY:
The study aims to develop a novel brief motivational mobile health (mHealth) intervention for frequent and/or high-intensity cannabis use for non-collegiate young adults. A total of 120 young adults (ages 18-29, not enrolled at or attending a 4-year college or university) will be randomized to receive a mHealth intervention with text messages for five weeks or to an online resource/program with psychoeducation information about cannabis. The mHealth intervention will focus on prompting the young adult to reflect on their journey with cannabis and to reflect on their personal goals and how cannabis is reflected in these goals. Additional mini-modules are included related to topics such as motivations for use, perceived norms and tracking cannabis use. Participants will return to the program each week to reflect on the prior week and reflect on goals for the upcoming week. All participants will complete a program satisfaction survey and complete follow-up assessments at 3- and 6-months post-program.

ELIGIBILITY:
Inclusion Criteria:

* 18-29 years old
* reside in Washington State
* have valid email address
* report using cannabis on 15 or more days in the past month, and/or using high THC concentration products in the past month (>60% THC)
* have a mobile phone and agree to receive text messages and has an internet browser
* not attending or enrolled at a 4-year college or university or graduate/professional school.

Exclusion Criteria:

* females who are pregnant or trying to become pregnant
* those who are in substance abuse treatment at screening
* those attending or enrolled at a 4-year college or university or graduate/professional school.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Cannabis use - typical hours high in a week | Baseline, 3-month follow-up, 6-month follow-up
  The count of the self-reported typical number of hours high per week during the past month
Negative cannabis-related consequences | Baseline, 3-month follow-up, 6-month follow-up
  Total sum score on the Marijuana Consequences Checklist based on number of self-reported cannabis-related consequences experienced in the past month. Higher scores indicate reporting greater number of negative cannabis-related consequences.

SECONDARY OUTCOMES:
Cannabis use - Number of sessions | Baseline, 3-month follow-up, 6-month follow-up
  Self-reported number of times/sessions used cannabis on the typical day during the past month

CONTACTS AND LOCATIONS:
Overall Officials: Christine M Lee, PhD, Principal Investigator — leecm@uw.edu
Locations (1):
- University of Washington, Seattle, Washington, United States